CLINICAL TRIAL: NCT02106650
Title: A Phase 2, Single-Arm, Open-Label, Multicenter, Study of Folotyn® (Pralatrexate Injection) in Combination With Oral Leucovorin to Prevent or Reduce Mucositis in Patients With Hematological Malignancies Including PTCL and CTCL
Brief Title: Phase II Study of Folotyn With Leucovorin to Prevent/Reduce Mucositis in Patients With Hematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Collaborators: Axis Clinicals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SPI-FOL-14-201
Record Dates: First submitted 2014-03-28; First posted 2014-04-08 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Relapsed Peripheral T-Cell Lymphoma; Refractory Peripheral T-Cell Lymphoma
Keywords: Relapsed PTCL; Refractory PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — 10-propargyl-10-deazaaminopterin; Leucovorin; Folic Acid; Vitamin B 12

ARMS (1):
- Folotyn and Leucovorin (Experimental): Folotyn will be administered by IV push at a dose of 30 mg/m2 once weekly for 6 weeks in each cycle, followed by 1 week of rest (no treatment).
  Leucovorin (25 mg tablets) will be taken orally tid for 2 days for a total of six doses (150 mg cumulative weekly dose), beginning 24 hours after each dose of Folotyn is administered.
  Folic acid and Vitamin B12 is given prior to initiation of Folotyn.
  Interventions: Drug: Folotyn and Leucovorin; Drug: Folic Acid; Drug: Vitamin B12

INTERVENTIONS:
Drug: Folotyn and Leucovorin
  Other Names: Pralatrexate (Folotyn)
Drug: Folic Acid — Folic acid (1.0 mg PO QD) is to be initiated at least 10 days prior to Folotyn administration, or per the USPI for Folotyn.
Drug: Vitamin B12 — Vitamin B12 (1 mg IM) is to be administered within 10 weeks prior to initiation of Folotyn and can be administered during Screening. Subsequent vitamin B12 injections may be given the same day as treatment with Folotyn and patients are to receive vitamin B12 every 8 to 10 weeks while treated with Folotyn.

SUMMARY:
This study is to evaluate the effect of leucovorin in preventing or reducing Folotyn-related Grade 2 or higher oral mucositis.

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, open-label, multicenter study to determine the effect of leucovorin in preventing or reducing Folotyn-related Grade 2 or higher oral mucositis in patients with hematological malignancies including PTCL and CTCL.

Patients with hematological malignancies, including PTCL and CTCL, will be enrolled based on meeting all protocol eligibility criteria. The primary endpoint will be evaluated in the first 7-week treatment cycle. For patients who respond to study treatment, the Investigator can treat patients for a total of 6 cycles. Approximately 37 patients will be enrolled. Safety, as assessed by reported SAEs, will continue to be monitored during the optional treatment period. Efficacy will be followed to the extent that it is evaluated according to the Institution's standard of care. No formal analysis of efficacy will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is diagnosed with hematological malignancies including PTCL and CTCL and are eligible for treatment with a dose of 30 mg/m^2
2. Patient is at least 18 years of age
3. Patient has been informed of the investigational nature of this study and has given written Informed Consent and is able to adhere to dosing and visit schedules and meet all study requirements
4. Patient has recovered from the toxic effects of prior therapy, and is at least 30 days from the most recent cytotoxic therapy, prior to enrollment
5. Patient has adequate hematologic, hepatic, and renal function as defined by:

   * ANC ≥1000/µL
   * Platelet count ≥100,000/µL
   * Total bilirubin ≤1.5 mg/dL
   * Aspartate aminotransferase/serum glutamic-oxaloacetic transaminase (AST/SGOT), alanine aminotransferase/serum glutamic-pyruvic transaminase (ALT/SGPT), and gamma-glutamyltransferase (GGT) ≤2.5 xupper limit of normal (ULN) (AST/ALT/GGT ≤5 xULN if documented hepatic involvement with lymphoma)
   * Creatinine ≤2.0 mg/dL or calculated creatinine clearance ≥50 mL/min
6. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤2
7. Females of childbearing potential are to agree to practice a medically acceptable contraceptive regimen (including a barrier method) from study treatment initiation until at least 30 days after the last administration of Folotyn or leucovorin, whichever is last, and are to have a negative urine beta human chorionic gonadotropin (β-HCG) pregnancy test within 14 days prior to the first day of study treatment. Females who are postmenopausal for at least 1 year (defined as >12 months since last menses) or are surgically sterilized do not require this test
8. Male patients are to agree to use a barrier method of contraception from study treatment initiation until at least 90 days after the last administration of Folotyn

Exclusion Criteria:

1. Patient has congestive heart failure Class III/IV according to the New York Heart Association (NYHA) Functional Classification
2. Patient has uncontrolled hypertension
3. Patient has known, uncontrolled human immunodeficiency virus (HIV)-positive diagnosis
4. Patient has symptomatic central nervous system (CNS) metastases or lesions for which treatment is required. Patients who received prophylactic CNS treatment are eligible
5. Patient has an active uncontrolled infection, underlying medical condition, or other serious illness that would impair the ability of the patient to receive protocol treatment
6. Patient has had major surgery within 14 days prior to enrollment
7. Patient has used any investigational drugs, biologics, or devices within 14 days prior to study treatment or plans to use any of these during the course of the study
8. Patient has had previous exposure to Folotyn within 6 months of study enrollment
9. Patient is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Grade 2 Oral Mucositis Prevention | 15 weeks
  To evaluate the effect of leucovorin in preventing or reducing Folotyn-related Grade 2 or higher oral mucositis.

SECONDARY OUTCOMES:
Grade 3 Oral Mucositis Prevention | 15 weeks
  To evaluate the effect of leucovorin in preventing or reducing Folotyn-related Grade 3 or higher oral mucositis.
Grade 2 Oral Mucositis Duration of first occurrence | 15 weeks
  To evaluate the time to first occurrence of Folotyn-related Grade 2 or higher oral mucositis.
Grade 2 Oral Mucositis Duration | 15 weeks
  To evaluate the duration of Folotyn-related Grade 2 or higher oral mucositis.
Effectiveness of Leucovorin in Folotyn dose modification | 15 weeks
  To evaluate the effect of leucovorin on the number and proportion of patients whose subsequent dose of Folotyn is omitted, delayed, or reduced due to the onset of oral mucositis.
Objective Response Rate | 17 weeks
  To evaluate objective response rate (ORR) of Folotyn in patients with relapsed or refractory (R/R) PTCL.

CONTACTS AND LOCATIONS:
Overall Officials: Wasim Khan, MD, Study Director — Acrotech Biopharma Inc.
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Cancer Center of Kansas, Wichita, Kansas
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Iyer SP, Dakhil S, Shinohara MM, Zain J, Acosta M, Foss F. Pralatrexate injection combined with oral leucovorin for mucositis management in PTCL/CTCL treatment: a multicenter phase 2 trial. Blood Neoplasia. 2024 Nov 2;2(1):100055. doi: 10.1016/j.bneo.2024.100055. eCollection 2025 Feb. PMID 40546726